CLINICAL TRIAL: NCT06022419
Title: Conservative Therapy of Proximal Phalanx Fractures - a Prospective Randomized Study Comparing the Lucerne Cast With Finger Splinting
Brief Title: Conservative Therapy of Proximal Phalanx Fractures - Comparing the Lucerne Cast With Finger Splinting
Acronym: LuCa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Paul L Hoppe, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1526/2023
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Proximal Phalanx Fracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lucerne Cast (Active Comparator)
  Interventions: Procedure: Lucerne Cast
- Forearm Cast and Finger Splint (Active Comparator)
  Interventions: Procedure: Forearm Cast and Finger Splint

INTERVENTIONS:
Procedure: Lucerne Cast — Patients receiving reduction of fractured finger and subsequent customization of a lucerne cast. Duration of cast treatment is determined with 4 weeks.
  Arms: Lucerne Cast
Procedure: Forearm Cast and Finger Splint — Patients receiving reduction of fractured finger and subsequent customization of a forearm cast with a finger splint. Duration of cast treatment is determined with 4 weeks.
  Arms: Forearm Cast and Finger Splint

SUMMARY:
The purpose of this prospective randomized controlled clinical trial is to evaluate if the lucerne cast leads to a better functional outcome than a forearm cast with a finger splint in patients with a proximal phalanx fracture.

DETAILED DESCRIPTION:
This study represents a prospective randomized controlled clinical trial comparing two different conservative treatment options in patients with proximal phalanx fractures.

Patients meeting the inclusion criteria will be enrolled in the present study provided they give their consent. Informed written consent will be obtained. Randomization will be performed according to the CONSORT Guidelines of Prospective Randomized Trials using the software "Randomizer" by the Medical University of Graz. Patients allocated to the control group will receive a forearm cast with a finger splint, while patients in the study group will receive the lucerne cast. Both groups will receive the allocated cast for 4 weeks. Clinical outcome will be assessed 12 weeks after trauma.

ELIGIBILITY:
Inclusion Criteria:

* Proximal phalanx fracture in the fingers (II - V)
* Patient age between 18 and 70 years

Exclusion Criteria:

* Condylar fracture
* Avulsions of the collateral ligament
* Pathologic fracture
* Intraarticular fracture
* Patients unable to consent
* Polytraumatized patients
* Patients initially presenting more than 7 days after injury
* Pregnancy
* Compound fractures
* Multiple hand injuries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Brief Michigan-Hand-Outcome-Questionnaire | at 12 weeks
  patient-based standardised questionnaire (12 items, range 0-100, 100=ideal function, 0=poorest function)

SECONDARY OUTCOMES:
Treatment Failure | at 1, 2, 4 and 12 weeks
  Occurrence of indication for surgery (malrotation, axial deviation >10°, dorsal angulation >20°) after primary reposition

OTHER OUTCOMES:
Visual Analogue Scale (VAS) | at 0, 1, 2, 4 and 12 weeks
  Pain evaluation on a psychometric response scale (range 0-10, 0=no pain, 10=maximum pain)
Strength Measurement | at 4 and 12 weeks
  dynamometer-based strength evaluation
Range of Motion (ROM) Assessment | at 4 and 12 weeks
  goniometer-based ROM evaluation of hand and wrist
Delayed Bone Healing | at 12 weeks
  number of participants with bone non-union at end of study
Radiological Outcome | at 0, 1, 2, 4 and 12 weeks
  x-ray based outcome of fracture healing in terms of axial deviation (measured in °)
Radiological Outcome | at 0, 1, 2, 4 and 12 weeks
  x-ray based outcome of fracture healing in terms of length deviation and dislocation (measured in mm)
Quick DASH-Score | at 0, 1, 2, 4 and 12 weeks
  patient-based standardised questionnaire (11 items, range 0-100, 100=ideal function, 0=poorest function)
Brief Michigan-Hand-Outcome-Questionnaire | at 0, 1, 2 and 4 weeks
  patient-based standardised questionnaire (12 items, range 0-100, 100=ideal function, 0=poorest function)
Occurrence of Complications | at 0, 1, 2, 4 and 12 weeks
  Occurrence of complications due to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerhild Thalhammer, M.D., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna - Department of Orthopedics and Trauma-Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No